CLINICAL TRIAL: NCT01386411
Title: Understanding Decision Making Processes for Undergoing Genetic Testing Among Women With Newly Diagnosed Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-086
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: Genetic testing; BRCA testing; Ashkenazi descent; 11-086
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood leucocytes and/or mouthwash-collected buccal epithelial cells)

GROUPS / COHORTS (1):
- Women with Breast Cancer: The proposed investigation is a prospective cohort study. Women with newly diagnosed breast cancer will decide whether to undergo BRCA testing either before or after completion of local surgical treatment.
  Interventions: Genetic: BRCA testing and questionnaire assessments

INTERVENTIONS:
Genetic: BRCA testing and questionnaire assessments — If they consent to enroll, they will complete an instrument evaluating their beliefs regarding the value of genetic testing (Assessment 1). After that, they will decide whether they wish to attend an information session on genetic predisposition. If they do, after completing that information session they will complete a follow-up instrument (Assessment 2), and will then decide to either immediately donate a sample for immediate testing, or to defer the decision until after surgery. Women will be given the results of their genetic testing in the context of a standard results counseling session, after which they will continue with clinical care. They will be followed for clinical decision, especially whether or not they undergo CPM.

SUMMARY:
Genes are the "blueprints" for our bodies. Some people are born with an abnormal copy ("mutation") of a gene. These people may have a higher chance of getting a disease. Different mutations in different genes cause different diseases. Some women get breast cancer because they are born with an abnormal copy of a gene called BRCA1 or BRCA2. These women also have a higher chance of getting ovary cancer. Women with breast cancer and an abnormal copy of BRCA1 or BRCA2 also have a higher chance of getting a second breast cancer in their other breast. Because of this, women who might have a mutation may have genetic testing soon after their breast cancer diagnosis to learn about their risks of getting another cancer.

Genetic testing may be done right after a woman has been diagnosed with breast cancer. It may also be done later, after surgery is done to treat the cancer. The investigators do not know when it is best to do genetic testing. The investigators are doing this study to try to understand whether women prefer testing before or after surgery. The investigator also want to find out how they feel about their choice later on, when their diagnosis in more in their past.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer or DCIS
* Appropriate for genetic testing, defined as if they meeting one or more of the following criteria (note that patients may be appropriate for genetic testing even if they do not meet these criteria, but NCCN and most payers recognize these groups as clearly appropriate for testing)
* Must be a primary malignancy (not recurrence), but can be second diagnosis if is a contralateral cancer and the first cancer was not treated with mastectomy
* Female age ≥18,
* If Ashkenazi Jewish: Breast cancer diagnosis ≤ 60. Subjects will be presumed to be of Ashkenazi ethnicity if Jewish religious preference is confirmed in subject and at least 1 parent, unless they explicitly endorse Sephardic, Iranian, Yemeni/Ethiopian, or Bukharan Jewish Decent, in which case non-Ashkenazi criteria will be applied.

If not Ashkenazi Jewish:

* Breast cancer diagnosis ≤ 45 OR
* Bilateral breast cancer, with first diagnosed ≤ 50 OR
* Breast cancer diagnosed at any age with a male relative with breast cancer OR
* Breast cancer diagnosis ≤ 50 with one or more of the following::

  * 1 or more relative with breast cancer ≤ 50 or
  * 1 or more relative with ovarian cancer
* Have not completed definitive surgical treatment
* For patients planning mastectomy for treatment, has not yet undergone mastectomy
* For patients planning breast conservation for treatment, has not yet begun adjuvant radiation therapy

Exclusion Criteria:

* LCIS without invasive cancer (IDC or ILC) and without DCIS
* Previous breast cancer treated with mastectomy
* Plan for neoadjuvant chemotherapy before surgery
* Unable to complete English language questionnaires, as instruments have not been validated in non-English speaking populations

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a prospective study of women who meet a subset of the NCCN criteria for genetic testing and are presenting to the Breast Surgery Clinic for treatment of a newly diagnosed breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
To determine the relative proportions of women offered genetic testing after a breast cancer diagnosis who decide to have BRCA testing | 2 years
  Either before completing definitive local surgical treatment (pre-surgical testing), after definitive surgical treatment (post-surgical) Women will be evaluated for their levels of general and cancer specific distress, coping style, and stage of decision-making with respect to PM (as this is the primary clinical reason for undergoing immediate testing).

SECONDARY OUTCOMES:
To determine the relative proportions of women who decide to undergo prophylactic mastectomy (PM) | 2 years
  The decision-making on prophylactic mastectomy (PM) will be obtained from the immediate and delayed BRCA genetic testers at Assessment 3. This will be a binary outcome of PM vs. no PM.
To assess the factors associated with the decision to choose pre- or post surgical testing. | 2 years
  We will compare the BRCA genetic testers (pooling immediate and delayed to boost the sample size) and the decliners on the summary scores of several psychosocial assessments using independent-sample t-tests for continuous variables (e.g., distress as measured by the BSI and IES) and non-parametric tests for categorical variables such as exact binomial test, Fisher's exact test, or the Chi-square test as appropriate (e.g., the blunters vs. monitors dichotomization) .

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm